CLINICAL TRIAL: NCT05970354
Title: Lidocaine-Prilocaine Cream as Analgesic for Outpatient Gynecological Procedures; A Randomized-Control Trial
Brief Title: EMLA Cream as Analgesic for Outpatient Gynecological Procedures
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: CAMC Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 22-910
Record Dates: First submitted 2023-07-07; First posted 2023-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Pain
Keywords: intra-uterine device insertion; hysteroscopy; endometrial biopsy
MeSH Terms: conditions — Pain | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- EMLA Cream (Active Comparator): 5 grams will be applied to patient's cervix 7 minutes before gynecological procedure
  Interventions: Drug: EMLA Cream
- VersaPro Cream (Placebo Comparator): 5 grams will be applied to patient's cervix 7 minutes before gynecological procedure
  Interventions: Drug: VersaPro Cream Base for Compounding

INTERVENTIONS:
Drug: EMLA Cream — Eutectic Mixture of Local Anesthetics (Lidocaine 2.5% and Prilocaine 2.5%)
  Arms: EMLA Cream
Drug: VersaPro Cream Base for Compounding — Placebo
  Arms: VersaPro Cream

SUMMARY:
The goal of this clinical trial is to compare pain perception in the study participant population undergoing the following gynecological procedures: Intra Uterine Device (IUD) insertion, hysteroscopy, and endometrial biopsy and given either Eutectic Mixture of Local Anesthetics (EMLA) cream or a placebo. The main question to answer is:

• Does EMLA cream reduce pain when administered during the following gynecological procedures: IUD insertion, hysteroscopy, and endometrial biopsy?

Participants will be asked to do assess their pain on the Visual Analogue Scale through 3 times during the procedure. Researchers will compare the study group with those receiving placebo group to see if there is a difference in pain scores.

DETAILED DESCRIPTION:
Gynecologic outpatient procedures such as intra-uterine device (IUD) insertion, hysteroscopy and endometrial biopsies (EMB) have no standard of care for pain management. This has resulted in acute pain for patients. One local anesthetic, Eutectic Mixture of Local Anesthetics (EMLA) cream (Lidocaine 2.5%/Prilocaine 2.5%), has shown to decrease perceived pain during hysteroscopy and IUD placement when compared to a placebo. The purpose of this study is to evaluate whether EMLA cream reduces pain during the following outpatient procedures: EMB, hysteroscopy, and IUD placement. Through a randomized control double-blind trial, study participants will have either 5 grams of EMLA cream or 5 grams of placebo applied to their cervix 7 minutes prior to the procedure. Patients' intensity of pain will be assessed using the Visual Analogue Scale (VAS) immediately after speculum placement, during the procedure, and immediately after completion of the procedure. Pain scores will be compared between the study and placebo group.

ELIGIBILITY:
Inclusion Criteria:

* Patient will undergo one of the following procedures: intra-uterine device insertion, hysteroscopy, or endometrial biopsies

Exclusion Criteria:

* Known hypersensitivity to amide anesthetics
* Pre-existing methemoglobinemia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Visual Analogue Scale Pain Score 1 | At time of speculum placement for procedure
  Scale of 0-10 on a self-reported pain score
Visual Analogue Scale Pain Score 2 | At start of cervical manipulation
  Scale of 0-10 on a self-reported pain score
Visual Analogue Scale Pain Score 3 | 2 minutes after speculum removal
  Scale of 0-10 on a self-reported pain score

CONTACTS AND LOCATIONS:
Overall Officials: Alex Poulsen, DO, Principal Investigator — West Virginia School of Medicine--Charleston Division
Locations (1):
- Charleston Area Medical Center Institute for Academic Medicine, Charleston, West Virginia, United States